CLINICAL TRIAL: NCT06341491
Title: The Study of Delay Discounting Propensity Among Beneficiaries of the Pé-de-Meia Program: The High School Savings Plan
Brief Title: The Study of Delay Discounting Among Beneficiaries of the Pé-de-Meia Program
Status: Not yet recruiting | Type: Observational
Sponsor: Federal Institute of Education, Science and Technology of the State of Mato Grosso (Other)
Responsible Party: Principal Investigator, Pamela Rodrigues Miranda, PROFESSOR, Federal Institute of Education, Science and Technology of the State of Mato Grosso
Other Study IDs: obs. Delay Discounting
Record Dates: First submitted 2024-03-15; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Delay Discounting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants of the Pé-de-Meia Program
  Interventions: Behavioral: Pé-de-Meia Program

INTERVENTIONS:
Behavioral: Pé-de-Meia Program — The "Pé-de-Meia" Program was established by the Brazilian Federal Government with the aim of encouraging the retention of low-income students in high school by providing maintenance scholarships and savings opportunities. To be eligible for the program, a young person must: Be properly enrolled in a regular public high school course, be between 14 to 24 years old, come from a low-income family, and be registered in the Bolsa Família Program. The Program offers four types of incentives:
  An enrollment grant registered at the beginning of the academic year, paid once a year in the amount of 200 BRL.
  A minimum school attendance of 80% of the total class hours, paid in nine installments throughout the year at 200 BRL each.
  Proven participation in the National High School Exam (ENEM), paid once to the student enrolled in the third year of high school, in the amount of 200 BRL.
  Completion of the high school academic years, paid in a single installment of 1,000 BRL.

SUMMARY:
The aim of this observational study is to explore how the "Pé-de-Meia" Program, a policy of the Brazilian Federal Government designed to encourage the retention and completion of studies by students from low-income families, affects both the students' tendency towards delay discounting and their academic performance. The study seeks to answer the following questions:

How does the "Pé-de-Meia" Program affect the students' propensity for delay discounting? Is there a relationship between the level of delay discounting among students, their academic performance, and school attendance? Participants in the study, high school students enrolled in the "Pé-de-Meia" Program, will undergo assessments to measure their level of delay discounting. The academic performance and school attendance of the participants will be monitored and analyzed in relation to their propensity for delay discounting

ELIGIBILITY:
Inclusion Criteria:

High school students, Students from public schools; Students from low-income families. -

Exclusion Criteria:

Students with a formal psychological report; students with a formal psychiatric report.

-

Ages: 14 Years to 24 Years | Sex: All
Age Groups: Child, Adult
Study Population: Youth between 14 and 24 years of age, duly enrolled in public education institutions and belonging to families that benefit from the Bolsa Família Program.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Delay discounting | April 2024, July 2024, October 2024, December 2024, February 2025, April 2025, July 2025, October 2025, December 2025
  Delay discounting measured by the Monetary Choice Questionnaire (MCQ).0.0 indicates an absence of discounting, meaning the individual values immediate and future rewards equally. This can be interpreted as a preference for delayed rewards or a long-term perspective.
  0.5 indicates strong discounting, meaning the individual significantly devalues future rewards in favor of immediate ones. This is seen as an indication of high impulsivity.
Academic performance - grades | December 2024 and December 2025
  Academic performance will be assessed based on school grades, categorized as follows: grades below 6 will indicate low performance; grades between 6 and 8 will reflect a medium performance; and grades between 8 and 10, a high performance
School attendance | December 2024 and December 2025
  School attendance will be evaluated based on the regularity of class attendance, organized into the following categories: an attendance rate below 80% will be considered low, while an attendance rate of 80% or more will indicate excellent school attendance.

IPD SHARING:
Plan to Share IPD: Undecided
I will review every request and make a decision later.